CLINICAL TRIAL: NCT04363359
Title: Immunogenicity and Safety of Quadrivalent Influenza Vaccine In 6 to 35 Months Population: a Randomized, Double-blind, Parallel-group Ⅱ Phase of Clinical Trials
Brief Title: Clinical Trial of Quadrivalent Influenza Virus Split Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CXSL1900048-Ⅰ+Ⅱ
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quadrivalent influenza vaccine HD (Experimental): Participants randomized to receive two injections of 0.5 mL quadrivalent influenza vaccine at Day 0 and 28.
  Interventions: Biological: 0.5ml Quadrivalent influenza vaccine
- Quadrivalent influenza vaccine LD (Experimental): Participants randomized to receive two injections of 0.25 mL quadrivalent influenza vaccine at Day 0 and 28.
  Interventions: Biological: 0.25ml Quadrivalent influenza vaccine
- Trivalent influenza vaccine Victoria (Active Comparator): Participants randomized to receive two injections of 0.25 mL trivalent influenza vaccine containing B/Victoria strain at Day 0 and 28.
  Interventions: Biological: 0.25ml Trivalent influenza vaccine(B/V)
- Trivalent influenza vaccine Yamagata (Active Comparator): Participants randomized to receive two injections of 0.25 mL trivalent influenza vaccine containing B/Yamagata strain at Day 0 and 28.
  Interventions: Biological: 0.25ml Trivalent influenza vaccine(B/Y)

INTERVENTIONS:
Biological: 0.5ml Quadrivalent influenza vaccine — The inactivated split virion vaccines contained 15 μg of each hemagglutinin antigen of influenza A/H1N1, A/H3N2, B/Victoria and B/Yamagata strains
  Arms: Quadrivalent influenza vaccine HD
Biological: 0.25ml Quadrivalent influenza vaccine — The inactivated split virion vaccines contained 7.5 μg of each hemagglutinin antigen of influenza A/H1N1, A/H3N2, B/Victoria and B/Yamagata strains
  Arms: Quadrivalent influenza vaccine LD
Biological: 0.25ml Trivalent influenza vaccine(B/V) — The inactivated split virion vaccines contained 7.5 μg of each hemagglutinin antigen of influenza A/H1N1, A/H3N2 and B/Victoria strains
  Arms: Trivalent influenza vaccine Victoria
Biological: 0.25ml Trivalent influenza vaccine(B/Y) — The inactivated split virion vaccines contained 7.5 μg of each hemagglutinin antigen of influenza A/H1N1, A/H3N2 and B/Yamagata strains
  Arms: Trivalent influenza vaccine Yamagata

SUMMARY:
To evaluate the immunogenicity and safety of 2 doses of quadrivalent influenza virus split vaccine in healthy population aged 6-35 month., so as to provide a data support for phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 6-35 months.
* Volunteer legal guardian or client informed consent, voluntarily participate in and sign informed consent.
* The volunteer legal guardian or client has the ability (non-illiterate) to understand the study procedures, to use a thermometer, scale, and fill in a diary card as required, and be able to complete the clinical study in compliance with the clinical trial protocol.

Exclusion Criteria:

* The underarm body temperature on the day of enrollment was > 37.0℃.
* Have been suffering from influenza within the previous 3 months (confirmed by either clinical, serological or microbiological methods).
* Any previous influenza vaccination (registered or experimental) within 6 months or any planned influenza vaccination during the study period.
* Allergic to any component of the vaccine, a history of allergic reactions to eggs or gentamicin sulfate.
* A history of severe allergy to any vaccine or drug.
* Preterm birth (delivered before 37 weeks of gestation), low birth weight baby (birth weight < 2300g for girls, <2500g for boys).
* Dystocia, asphyxia rescue, nervous system damage history;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Acute illness, severe chronic illness or acute attack of chronic disease on the day of vaccination;
* A history of live attenuated vaccination within 14 days prior to vaccination and a history of other vaccinations within 7 days prior to vaccination;
* Patients who received immunoenhancement or inhibitor therapy within 3 months (continued oral or intravenous administration for more than 14 days);
* Congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* History of asthma, past two years of instability requiring emergency treatment, hospitalization, intubation, oral or intravenous administration of corticosteroids;
* Have received blood or blood-related products;
* A history of convulsion, epilepsy, encephalopathy, guillain-barre syndrome, a history of mental illness or a family history;
* A history of abnormal coagulation function (such as coagulation factor deficiency, coagulation disease);
* Planning to relocate before the end of the study or to leave for an extended -period during the scheduled study visit;
* Participating in or planning to participate in other clinical trials in the near future;
* The investigators determined that any conditions were inappropriate to participate in the clinical trial.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 1980 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
seroconversion rate of HI antibodies | 56 days
  28 days after receiving two doses of vaccine in subjects aged 6-35 months, seroconversion rate of HI antibodies against any subtype of influenza virus in each group.
seroprotection rate of HI antibodies | 56 days
  28 days after receiving two doses of vaccine in subjects aged 6-35 months, seroprotection rate of HI antibodies against any subtype of influenza virus in each group.
GMT and GMI of HI antibodies | 56 days
  28 days after receiving two doses of vaccine in subjects aged 6-35 months, GMT and GMI of HI antibodies against any subtype of influenza virus in each group.

SECONDARY OUTCOMES:
Reactogenicity Events | 30 days and 6 months
  1. The proportion of all adverse reactions/events in each group through 30 days after the second dose.
  2. The proportion of serious adverse events (SAE) within 6 months after inoculation in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Shilei Wang, PhD, Principal Investigator — Shanghai Institute Of Biological Products
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04363359/Prot_SAP_000.pdf